CLINICAL TRIAL: NCT00453193
Title: A Phase II Study of Alemtuzumab and Pentostatin In T-Cell Neoplasms
Brief Title: Alemtuzumab and Pentostatin In T-cell Neoplasms
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0408
Record Dates: First submitted 2007-03-26; First posted 2007-03-28 (Estimated); Results first posted 2011-03-28 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Lymphoma; Leukemia
Keywords: T-Cell Neoplasms; Alemtuzumab; Pentostatin; Campath-1H; Deoxycoformycin; Lymphoma; Leukemia
MeSH Terms: conditions — Lymphoma; Leukemia | interventions — Pentostatin; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alemtuzumab + Pentostatin (Experimental): Alemtuzumab 30 mg intravenous (IV) three times weekly; Pentostatin 4 mg/m^2 IV weekly for 4 weeks then every 2 weeks
  Interventions: Drug: Pentostatin; Drug: Alemtuzumab

INTERVENTIONS:
Drug: Pentostatin — 4 mg/m^2 IV weekly for 4 weeks then every 2 weeks
  Other Names: Nipent®
Drug: Alemtuzumab — 30 mg IV three times weekly
  Other Names: Campath; CAMPATH-1

SUMMARY:
The goal of this clinical research study is to learn if giving pentostatin with alemtuzumab can help to control T-cell malignancy. The safety of this combination therapy will also be studied.

DETAILED DESCRIPTION:
Alemtuzumab is an antibody protein that is directed towards a marker molecule on the surface of both B- and T- lymphoid cells. It is currently approved for use in treating patients with chronic lymphocytic leukemia and has been studied in treating patients with a number of T-cell malignancies. Alemtuzumab has been found to be effective in these conditions. Pentostatin is a drug that is approved for treating patients with hairy cell leukemia, a B-cell malignancy. Pentostatin has also been studied in a number of T-cell cancers and has been found to be effective. The purpose of this study is to see whether combining these drugs will prove to be more effective.

If you are found to be eligible to take part in this study, you will receive pentostatin through a central venous catheter in your vein once a week for 4 weeks and then every 2 weeks until the achievement of best response. A central venous catheter is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your physician will explain this procedure to you in more detail and you will be required to sign a separate consent form for this procedure.

Alemtuzumab will also be given through a vein catheter on Days 1, 2, and 3. The dose of alemtuzumab that you receive will be increased each day for the first 3 days to make sure that you tolerate it. It will then be given three times per week until you achieve the best response. If you develop reactions to alemtuzumab when given through a vein, you may receive it by injections of the same dose under the skin.

During the treatment, you will have blood (about 2 tablespoons) drawn once a week for the first 4 weeks for routine blood tests. These blood tests will then be repeated every 2 to 4 weeks for the remainder of the study. At the end of treatment a bone marrow examination will be repeated to document your response. Also, if you had a chest X-ray or CT scans, these will be repeated to confirm your level of response.

The maximum amount of time that alemtuzumab will be given is 3 months. The maximum amount of time that pentostatin will be given is 6 months. You may be able to receive the treatment will your local oncologists. However, you will have close follow-up at M. D. Anderson. You will be taken off this treatment if the disease gets worse during treatment or if unacceptable side effects develop.

You will be continued to be followed either directly or by telephone to evaluate your long-term response to treatment on this study.

This is an investigational study. Both alemtuzumab and pentostatin are commercially approved drugs that have been used to treat T-cell malignancies. A total of 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

This is an investigational study. Both alemtuzumab and pentostatin are commercially approved drugs that have been used to treat T-cell malignancies. A total of 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older
2. Diagnosis of T lymphoid malignancy established by peripheral blood, bone marrow or tissue (skin, lymph node or other) examination and using the standard criteria.
3. Patients with untreated T-cell-prolymphocytic leukemia (T-PLL), peripheral T-cell lymphoma, hepatosplenic T-cell lymphoma and NK/T cell lymphoma are eligible.
4. Patients with relapsed/refractory T-PLL, T-lineage acute lymphoblastic leukemia (T-ALL), Adult T-cell leukemia/lymphoma (ATLL), peripheral T-cell lymphoma, hepatosplenic T-cell lymphoma and NK/T cell lymphoma and other T-lymphoid malignancies are eligible. Patients who have had prior therapy with either alemtuzumab or pentostatin as single agents are eligible.
5. Willing to use adequate contraception for the entire duration of the study.
6. Performance status 0-2.
7. Creatinine less than or equal to 2.0 mg/dL and calculated creatinine clearance greater than 40
8. Bilirubin less than or equal to 3.0 mg/dL, transaminases (aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT)) less than 4 x upper limit of normal unless related to the disease.
9. Left ventricular ejection fraction greater than 30%.

Exclusion Criteria:

1. Unable or unwilling to sign the consent form.
2. Pregnant or lactating
3. Known to be HIV+
4. Active and uncontrolled infection as judged by treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Andersons website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 8/241/2004 to 5/12/2009. All patients registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: Of the 26 enrolled, only 24 patients were included in this study.
Period: Overall Study
Arm/Group | Alemtuzumab + Pentostatin
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alemtuzumab + Pentostatin
Number analyzed (Participants) | 24
Age Continuous [Median (Full Range); unit: years] | 57 [21 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective Responses are Complete or Partial Responses: Complete Response defined as disappearance of all evidence of disease detectable by morphology of peripheral blood and bone marrow and computer tomography scanning at the end of therapy, if indicated; and Partial Response as 50% or more reduction in detectable disease, but short of complete response, maintained for 1 month or at least 50% reduction of sum of the products of the diameter of all lesions for 1 month.
Time Frame: After a maximum of 6 months of therapy maintained for one month.
Population: Analysis was per protocol.
Measure: Number; unit: Participants
Arm/Group | Alemtuzumab + Pentostatin
Number analyzed (Participants) | 24
Participants
  Complete Response | 11
  Partial Response | 2

ADVERSE EVENTS:
Time Frame: 5 years 2 months
Arm/Group | Alemtuzumab + Pentostatin
Serious Adverse Events (participants affected / at risk) | 15/24
Other Adverse Events (participants affected / at risk) | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alemtuzumab + Pentostatin (N=24)
elevated asparatate aminotransferase (Hepatobiliary disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (4)
Death (General disorders) | 8 (8)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Neutropenic Fever (Infections and infestations) | 1 (1)
Subdural Hematoma (Blood and lymphatic system disorders) | 1 (1)
sinusitis (Infections and infestations) | 1 (1)
non neutropenic fever (Infections and infestations) | 1 (1)
Granulocytopenia (Blood and lymphatic system disorders) | 1 (1)
increased liver function (Hepatobiliary disorders) | 1 (1)
headache (Nervous system disorders) | 1 (1)
fever (General disorders) | 1 (1)
Epididymitis (Blood and lymphatic system disorders) | 1 (1)
viral infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alemtuzumab + Pentostatin (N=24)
Hives (General disorders) | 9 (9)
Edema (General disorders) | 3 (3)
fatugue (General disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 15 (15)
Hepatic (Hepatobiliary disorders) | 7 (7)
Ocular (Eye disorders) | 2 (2)
Pain (General disorders) | 7 (7)
Renal (Renal and urinary disorders) | 5 (5)
tumor lysis syndrome (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes